CLINICAL TRIAL: NCT01435161
Title: The Effect of Nifedipine Versus Telmisartan on Prevention of Atrial Fibrillation Recurrence in Hypertensive Patients With Paroxysmal Atrial Fibrillation by Intensive Lower Blood Pressure
Brief Title: Nifedipine vs Telmisartan on Prevention of Atrial Fibrillation (AF) Recurrence in Hypertensive Patients With AF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Chief, Dept. of Cardiology, the second affiliated hospital of Chongqing medical university, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NTP-AF
Record Dates: First submitted 2011-09-14; First posted 2011-09-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Atrial Fibrillation
Keywords: paroxysmal atrial fibrillation, hypertension
MeSH Terms: conditions — Atrial Fibrillation; Hypertension | interventions — Nifedipine; Antihypertensive Agents; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nifedipine (Active Comparator): Patients in arm 1 receive Nifedipine;
  Interventions: Drug: Nifedipine,
- Telmisartan (Active Comparator): Arm 2 receive telmisartan
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Nifedipine, — Nifedipine 30-60mg/day
  Other Names: anti-hypertensive drugs, Atrial fibrillation
  Arms: Nifedipine
Drug: Telmisartan — Telmisartan 80-160mg/day
  Other Names: anti-hypertensive drugs, atrial fibrillation
  Arms: Telmisartan

SUMMARY:
Different lowing blood pressure strategies have a different clinical efficacies. Blocking the angiotensin II type 1 receptor (Telmisartan) reduces the incidence of episodes of atrial fibrillation in hypertensive patients with paroxysmal atrial fibrillation during 24 months than 30% compared to Nifedipine( Adalat GITS ).

A total of 160 subjects will be included in two study groups. The Group 1 will receive 80-160mg Telmisartan per day, the remaining patients will receive Nifedipine ( Adalat GITS). Follow-up is 24 months. The conventional 12-lead ECG recordings at twice weeks interval and 24hrs holter monitor will determine the cardiac rhythm and asymptomatic episodes of atrial fibrillation. The target of Blood pressure after 3 months is less than 130/80mmHg. Concomitant therapy with B-blocker and acethydrazide are allowed for the target blood pressure during the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented hypertensive patients with paroxysmal atrial fibrillation: ECG documentation of atrial fibrillation at least in one ECG recorded during the last 2 months prior to randomization plus additional ECG recording of sinus rhythm at least 12 hours after the above mentioned ECG documentation.
* Patients with hypertensive history were at least 5 years. Systolic pressure > 140mmHg, < 190mmHg, Diastolic pressure > 85mmHg. < 110mmHg.
* 40 < Age < 65 years

Exclusion Criteria:

* Strong clinical evidence for therapy with AT II/ACE inhibitors before 3 months of screening
* Therapy with antiarrhythmic agents of class I or class III within the last month, therapy with amiodarone within the last 3 months
* Direct current (DC) cardioversion within the last 3 months
* Symptomatic bradycardia
* Implanted pacemaker or implanted cardioverter/defibrillator with any antitachycardiac algorithm in use
* Cardiac surgery or cardiac catheter ablation within the last 3 months
* Typical angina pectoris symptoms at rest or during exercise
* Known coronary artery disease with indication for intervention
* Valvular disease > II degree
* Left ventricular ejection fraction < 40%
* Diastolic blood pressure > 110mm Hg at rest
* Symptomatic arterial hypotension
* Known renal artery stenosis
* Serum creatinine > 1.8 mval/l
* Relevant hepatic or pulmonary disorders
* Hyperthyroidism manifested clinically and in laboratory
* Known drug intolerance for AT II inhibitors
* Females who are pregnant or breast feeding
* Females of childbearing potential who are not using a scientifically accepted method of contraception
* Participation in a clinical trial within the last 30 days
* Drug addiction or chronic alcohol abuse
* Legal incapacity, or other circumstances which would prevent the patient from understanding the aim, nature or extent of the clinical study
* Evidence of an uncooperative attitude

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Recurrence of Atrial Fibrillation | four years
  Recurrence of Atrial Fibrillation ( at least one readable conventional and Holter ECG recording)

CONTACTS AND LOCATIONS:
Overall Officials: Yuehui Yin, MD, Study Chair — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- 2ndChongqingMU, Chongqing, Chongqing Municipality, China